CLINICAL TRIAL: NCT02220504
Title: Clinical Outcome After Antipsychotic Treatment Discontinuation in Functionally Recovered First-episode Non-affective Psychosis Individuals: A 3-year Follow-up
Brief Title: 3-year Follow-up of Clinical Outcome After Antipsychotic Treatment Discontinuation in Psychosis Individuals
Acronym: ADARFEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Marques de Valdecilla (Other)
Collaborators: Centro de Investigación Biomédica en Red de Salud Mental (Network); Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, Benedicto Crespo-Facorro, Associate Professor of Psychiatry, Fundación Marques de Valdecilla
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADARFEP
Record Dates: First submitted 2014-08-13; First posted 2014-08-20 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Schizophrenia; Schizophrenia Relapse; Schizophrenia Spectrum and Other Psychotic Disorders
Keywords: Treatment; Maintenance
MeSH Terms: conditions — Schizophrenia; Schizophrenia Spectrum and Other Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Antipsychotic treatment discontinuation (DT)
  Interventions: Other: Antipsychotic treatment discontinuation
- Control group (Active Comparator): Maintenance antipsychotic treatment (MT)
  Interventions: Other: Maintenance antipsychotic treatment

INTERVENTIONS:
Other: Antipsychotic treatment discontinuation — Withdrawal of antipsychotic medication to stabilized patients.
  Arms: Intervention group
Other: Maintenance antipsychotic treatment — Maintenance antipsychotic medication to stabilized patients.
  Arms: Control group

SUMMARY:
This open-label, non-randomized, prospective study will evaluate the risk of symptoms recurrence during the three years after antipsychotic discontinuation in a sample of functionally recovered first-episode patients with schizophrenia spectrum disorder.

ELIGIBILITY:
Inclusion Criteria:

* Individuals included in the First Episode Psychosis Clinical Program (PAFIP) at the University Hospital Marqués de Valdecilla (Santander, Spain).
* A minimum of 18 months on antipsychotic treatment.
* Meeting clinical remission criteria for at least the 12 months prior to inclusion.
* Meeting the functional recovery criteria for at least the 6 months prior to inclusion.
* Stabilized at the lowest effective doses for at least the 3 months prior to inclusion.

Exclusion Criteria:

* Meeting Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for drug dependence.
* Meeting DSM-IV criteria for mental retardation.
* Having a history of neurological disease or head injury.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2004-07 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Relapse rate. | At 3 years.
  The main outcome was the percentage of relapse/exacerbation in the two groups of patients, discontinuation and maintenance.

SECONDARY OUTCOMES:
Clinical psychopathology. | At 3 years.
  Clinical psychopathology differences between groups are evaluated by the mean change from the study intake to 3 years for the severity of Clinical Global Impression scale (CGI), Brief Psychiatric Rating Scale expanded version of 24 items (BPRS), Scale for the Assessment of Positive Symptoms (SAPS) and Scale for the Assessment of Negative Symptoms (SANS) total scores.
Time to relapse. | At 3 years.
  Time to relapse in the two groups of patients, discontinuation and maintenance.
Clinical functionality. | At 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Benedicto Crespo-Facorro, Professor, Principal Investigator — University Hospital Marqués de Valdecilla, IDIVAL, Department of Psychiatry, School of Medicine, University of Cantabria, Santander, Spain. CIBERSAM Centro Investigación Biomédica en Red Salud Mental, Madrid, Spain
Locations (1):
- University Hospital Marques de Valdecilla, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mayoral-van Son J, de la Foz VO, Martinez-Garcia O, Moreno T, Parrilla-Escobar M, Valdizan EM, Crespo-Facorro B. Clinical outcome after antipsychotic treatment discontinuation in functionally recovered first-episode nonaffective psychosis individuals: a 3-year naturalistic follow-up study. J Clin Psychiatry. 2016 Apr;77(4):492-500. doi: 10.4088/JCP.14m09540. PMID 26759992